CLINICAL TRIAL: NCT01215253
Title: Late Sodium Current Blockade in High-Risk ICD Patients
Brief Title: Ranolazine Implantable Cardioverter-Defibrillator Trial
Acronym: RAID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Wojciech Zareba, MD PhD, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U01HL096607 (NIH)
Record Dates: First submitted 2010-09-30; First posted 2010-10-06 (Estimated); Results first posted 2018-06-15 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Ischemic Cardiomyopathy; Nonischemic Cardiomyopathy; Heart Failure
Keywords: Sudden Death; Ranolazine; Heart failure; Ventricular tachycardia; Ventricular fibrillation; Implantable cardioverter-defibrillator
MeSH Terms: conditions — Heart Failure; Death, Sudden; Tachycardia, Ventricular; Ventricular Fibrillation | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: No

ARMS (2):
- Ranolazine (Active Comparator): At enrollment, patients will be randomized to ranolazine or placebo. In the active drug arm each patient will be started on a 500 mg twice a day dose for one week with subsequent increase to 1000 mg twice a day at end of first week. For patients on anti-arrhythmic therapy at the time of randomization, their ECG will be checked at end of first week on 500 mg dose and again at end of second week on 1000 mg dose. For patients with CrCl <60ml/min prior to randomization, their CrCl will be checked again at 2 weeks and study drug discontinued if <30ml/min. For patients with CrCl <60ml/min at 2 weeks, their CrCl will be checked again at 4 weeks and study drug discontinued if <30ml/min.
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): At enrollment, patients will be randomized to ranolazine or placebo. In the active drug arm each patient will be started on a 500 mg twice a day dose for one week with subsequent increase to 1000 mg twice a day at end of first week. For patients on anti-arrhythmic therapy at the time of randomization, their ECG will be checked at end of first week on 500 mg dose and again at end of second week on 1000 mg dose. For patients with CrCl <60ml/min prior to randomization, their CrCl will be checked again at 2 weeks and study drug discontinued if <30ml/min. For patients with CrCl <60ml/min at 2 weeks, their CrCl will be checked again at 4 weeks and study drug discontinued if <30ml/min.
  Interventions: Drug: Ranolazine

INTERVENTIONS:
Drug: Ranolazine — At enrollment, patients will be randomized to ranolazine or placebo. In the active drug arm each patient will be started on a 500 mg twice a day dose for one week with subsequent increase to 1000 mg twice a day at beginning of second week.
  Other Names: Ranexa

SUMMARY:
The purpose of the study is to see how effective a drug called ranolazine is in reducing the risk of ventricular arrhythmia and death in people with implantable cardioverter-defibrillators (ICDs). This drug will be used with standard medications that is routinely prescribed in enrolled patients.

DETAILED DESCRIPTION:
There are limited treatment options for patients at high risk of ventricular arrhythmic events. Beta-blockers alone do not provide enough protection, sotalol has limited effectiveness, and amiodarone although effective in some groups of patients is used infrequently due to its side effects and limitations of a long-term use. Ischemia and cardiomyopathies are associated with a sodium overload of myocardial cells. Late sodium current plays a pivotal role in this process. Sodium overload leads to calcium overload of myocardial cells with consequent increased vulnerability of myocardium to ventricular tachyarrhythmias as well as increased impairment of diastolic relaxation of myocardium thereby augmenting the risk of ischemia and myocardial damage.

Ranolazine is a novel drug with anti-ischemic and antiarrhythmic properties that uniquely blocks late sodium current, decreases intracellular calcium overload, and improves diastolic relaxation of the ventricles. The antiischemic and antiarrhythmic properties of ranolazine might decrease the likelihood of arrhythmic events and improve the clinical course of patients with ventricular arrhythmias.

We designed a randomized double-blind placebo-controlled clinical trial enrolling 1,440 high-risk ICD patients who will be treated with ranolazine or placebo in addition to optimal medical therapy to test the hypothesis that late sodium current blockade contributes to significant reduction in the risk of arrhythmic events or death in high-risk ICD/cardiac resynchronization therapy-D patients.

ELIGIBILITY:
Inclusion Criteria:

1,440 high-risk patients with ischemic/nonischemic cardiomyopathy who receive their ICDs as standard of care for primary or secondary prevention of mortality following approved indications for ICD therapy. High-risk patients will be defined as:

Secondary Prevention Patients Subjects with ischemic or nonischemic cardiomyopathy, qualified for or with existing ICD (or CRT-D) after documented VT/VF or cardiac arrest (secondary prevention of mortality). Secondary prevention subjects with existing implants are eligible regardless of when the implant was received (subjects could be recruited from outpatient clinics or from inpatient activity including during re-implant or other procedures).

Primary Prevention Patients

1. Patients with primary prevention indications for ischemic or non-ischemic cardiomyopathy with EF≤35%, with existing devices (ICD/CRT-D), regardless of when the device was implanted, who have experienced at least ONE episode of VT/VF appropriately treated with ICD therapy (ATP or shock) or had untreated NSVT lasting at least 10 beats with heart rate of at least 170 bpm, documented by electrogram of their implanted device.
2. Patients with ischemic or non-ischemic cardiomyopathy with EF≤35%, who have been implanted within the last 2 years (initial ICD/CRT-D implants, including upgrades from pacemakers) who have NOT experienced VT/VF treated with ICD therapy (ATP or shock), AND who have one of the following additional criteria: BUN≥26 mg/dl or QRS>120ms or Atrial Fibrillation or NSVT documented by ECG/Holter or >500 Ventricular Premature Beats (VPBs)documented in a 24-hour Holter.

   * Stable optimal pharmacologic therapy for the cardiac condition
   * Age: equal to 21 years without upper limit

Exclusion Criteria:

* Patient receiving first device with coronary artery bypass graft surgery within the last 3 calendar months prior to date consent obtained
* Patients receiving first device with percutaneous coronary intervention within the last 1 calendar month prior to date consent obtained
* Patient receiving first device with enzyme-positive myocardial infarction with the past 3 calendar months prior to date consent obtained
* Patient receiving first device with angiographic evidence of coronary disease who are candidates for coronary revascularization and are likely to undergo coronary artery bypass graft surgery or percutaneous coronary intervention in the foreseeable future
* Patient in NYHA Class IV
* Patients receiving prophylactic ablation of ventricular substrate
* Patients with preexisting QTc prolongation >550ms
* Patients on strong CYP3A inhibitors (including ketoconazole, itraconazole, clarithromycin, nefazodone, nelfinavir, ritonavir, indinavir and saquinavir and moderate CYP3A inhibitors, including, diltiazem, verapamil, aprepitant, erythromycin, fluconazole and grapefruit juice or grapefruit-containing products.
* Patients on CYP3A inducers such as rifampin, rifabutin, rifapentine, phenobarbital, phenytoin, carbamazepine and St.John's wort
* Patients with inherited arrhythmia disorders such as Brugada's, ARVD, LQTS or hypertrophic cardiomyopathy
* Patient who is pregnant or plans to become pregnant during the course of the trial (patients at child bearing age who use prescribed pharmaceutical contraceptives could be enrolled)
* Patient with irreversible brain damage from preexisting cerebral disease
* Patient with presence of any disease, other than the patient's cardiac disease, associated with a reduced likelihood of survival for the duration of the trial, e.g., cancer, uremia, liver failure, etc.
* Patient with chronic renal disease with creatinine >2.5 mg/dl or creatinine clearance <30 ml/min
* Patient participating in any other clinical trial
* Patient unwilling or unable to cooperate with the protocol
* Patient who lives at such a distance from the clinic that travel for follow-up visits would be unusually difficult
* Patient who does not anticipate being a resident of the area for the scheduled duration of the trial
* Patients who are decisionally impaired adults, those of questionable capacity, and those who cannot consent for themselves will not be recruited for this study.
* Patient unwilling to sign the consent for participation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2011-09; Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Zareba, MD PhD, Principal Investigator — University of Rochester
Locations (90):
- United States (83):
  - University of Arizona, Tucson, Arizona
  - Arkansas Cardiology, Little Rock, Arkansas
  - Sequoia Hospital, East Palo Alto, California
  - Good Samaritan Hospital, Los Angeles, California
  - Huntington Memorial Hospital, Pasadena, California
  - Regional Cardiology Associates, Sacramento, California
  - Delta Heart and Medical Clinic, Stockton, California
  - University of Colorado Health - MHS, Colorado Springs, Colorado
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Washington Electrophysiology/Cardiovascular Research Institute, Washington D.C., District of Columbia
  - Bay Area Cardiology Associates, P.A., Brandon, Florida
  - University of Florida/Cardiovascular Medicine, Gainesville, Florida
  - University of Florida Health Science Center at Jacksonville, Jacksonville, Florida
  - Watson Clincia Center for Research Inc., Lakeland, Florida
  - Florida Hospital, Orlando, Florida
  - Tallahassee Research Institute, Inc., Tallahassee, Florida
  - Georgia Health Sciences University, Augusta, Georgia
  - Georgia Arrhythmia Consultants, Macon, Georgia
  - University of Chicago Hospital, Chicago, Illinois
  - Peakview Research Center, Fort Wayne, Indiana
  - LaPorte Hospital, Hobart, Indiana
  - University of Iowa, Iowa City, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Louisiana State University Health Sciences Center- New Orleans, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - MedStar Southern Maryland Hospital Center, Clinton, Maryland
  - Tufts-New England Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Massachusetts-Worchester, Worcester, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - William Beaumont Hospital - Royal Oak, Royal Oak, Michigan
  - Michigan Heart, Ypsilanti, Michigan
  - St. Luke's Hospital Association of Duluth, Duluth, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri, Columbia, Missouri
  - Kansas City Heart Foundation, Kansas City, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Morristown Memorial Hospital- Gagnon Cardiovascular Institute, Morristown, New Jersey
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Weill Cornell Medical College/New York Presbyterian Hospital, New York, New York
  - St. Luke's-Roosevelt Hospital, New York, New York
  - Hudson Valley Heart Center, Poughkeepsie, New York
  - The Valley Hospital, Ridgewood, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center,, Stony Brook, New York
  - Durham VA Medical Center, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - The Lindner Center for Research & Education, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - The MetroHealth System - Heart and Vascular Dept., Cleveland, Ohio
  - The Toledo Hospital/Northwest Ohio Cardiology Consultants, Toledo, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Portland VA Medical Ctr, Portland, Oregon
  - Abington Medical Specialists, Abington, Pennsylvania
  - Doylestown Cardiology Associates - VIAA, Doylestown, Pennsylvania
  - Doylestown Health Cardiology/Central Bucks, Doylestown, Pennsylvania
  - Lancaster Heart & Stroke Foundation, Lancaster, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center-Presbyterian, Pittsburgh, Pennsylvania
  - VA Pittsburgh Healthcare Center, Pittsburgh, Pennsylvania
  - Lankenau Institute for Medical Research, Wynnewood, Pennsylvania
  - Brigham and Women's Cardiovascular Associates, Warwick, Rhode Island
  - The Stern Cardiovascular Center, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Cardiopulmonary Research Science and Technology Inst., Dallas, Texas
  - Medicus Alliance CRO, Inc, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
  - Cardiovascular Associates Ltd., Chesapeake, Virginia
  - Walter Reed NMMC, Portsmouth, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Kootenai Heart Clinics, LLC, Spokane, Washington
  - Cardiac Study Center, Tacoma, Washington
  - CAMC Institute, Charleston, West Virginia
  - Marshfield Clinic, Marshfield, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Wheaton Franciscan All Saints, Racine, Wisconsin
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Queen's University, Kingston, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - CHUS (Sherbrooke University), Sherbrooke, Quebec
  - IUCPQ, Québec

IPD SHARING:
Plan to Share IPD: No
The RAID PI and Steering Committee with investigators from enrolling sites have designed a series of secondary substudies that will be disseminated as abstracts and manuscripts. External proposal of analyses of the RAID trial data will be reviewed bye the Steering Committee and analyses will be conducted by the Data Coordinating Center (DCC) of the trial.

REFERENCES:
- [Derived] Krzowski B, Kutyifa V, Vloka M, Huang DT, Attari M, Aktas M, Shah AH, Musat D, Rosenthal L, McNitt S, Polonsky B, Schuger C, Natale A, Ziv O, Beck C, Daubert JP, Goldenberg I, Zareba W. Sex-Related Differences in Ventricular Tachyarrhythmia Events in Patients With Implantable Cardioverter-Defibrillator and Prior Ventricular Tachyarrhythmias. JACC Clin Electrophysiol. 2024 Feb;10(2):284-294. doi: 10.1016/j.jacep.2023.09.028. Epub 2023 Nov 29. PMID 38032582
- [Derived] Younis A, Goldenberg I, Farooq S, Yavin H, Daubert J, Raitt M, Mazur A, Huang DT, Mitchell BL, Rashtian MR, Winters S, Vloka M, Aktas M, Bernabei MA, Beck CA, McNitt S, Zareba W. Reduction in Ventricular Tachyarrhythmia Burden in Patients Enrolled in the RAID Trial. JACC Clin Electrophysiol. 2022 Jun;8(6):754-762. doi: 10.1016/j.jacep.2022.02.018. Epub 2022 Apr 27. PMID 35738852
- [Derived] Zareba W, Daubert JP, Beck CA, Huang DT, Alexis JD, Brown MW, Pyykkonen K, McNitt S, Oakes D, Feng C, Aktas MK, Ayala-Parades F, Baranchuk A, Dubuc M, Haigney M, Mazur A, McPherson CA, Mitchell LB, Natale A, Piccini JP, Raitt M, Rashtian MY, Schuger C, Winters S, Worley SJ, Ziv O, Moss AJ; RAID Trial Investigators. Ranolazine in High-Risk Patients With Implanted Cardioverter-Defibrillators: The RAID Trial. J Am Coll Cardiol. 2018 Aug 7;72(6):636-645. doi: 10.1016/j.jacc.2018.04.086. PMID 30071993

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1012 patients were recruited from 88 centers in the US and 7 centers in Canada
Period: Overall Study
Arm/Group | Ranolazine | Placebo
Started | 510 | 502
Completed | 424 | 439
Not Completed | 86 | 63
Not completed — Withdrawal by Subject | 57 | 35
Not completed — Physician Decision | 9 | 12
Not completed — Lost to Follow-up | 6 | 4
Not completed — Other | 14 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranolazine | Placebo | Total
Number analyzed (Participants) | 510 | 502 | 1012
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (10.3) | 64.2 (9.9) | 64.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 86 | 186
  Male | 410 | 416 | 826
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 12 | 29
  Not Hispanic or Latino | 493 | 490 | 983
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 85 | 85 | 170
  White | 404 | 410 | 814
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 12 | 2 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 31 | 31 | 62
  United States | 479 | 471 | 950

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Ventricular Tachycardia (VT) or Ventricular Fibrillation (VF) or Death
Description: Primary endpoint of the study will be defined as a composite endpoint consisting of Ventricular Tachycardia or Ventricular Fibrillation requiring antitachycardia pacing (ATP) therapy, implantable cardioverter-defibrillator (ICD) shock, or death, whichever occurs first.
Time Frame: 2 years of follow-up on average
Population: This outcome measure was an intent-to-treat analysis therefore all randomized subjects were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 510 | 502
Participants | 174 | 198
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority; p = 0.117, Regression, Cox; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.67 to 1.05]

2. Secondary Outcome: Number of Patients With VT or VF Requiring ICD Shock or Death
Description: Implantable cardioverter-defibrillator (ICD) shock for VT or VF or death, whichever occurs first.
Time Frame: 2 years of follow-up on average
Population: This outcome measure was an intent-to-treat analysis therefore all randomized subjects were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 510 | 502
Participants | 131 | 145
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority; p = 0.891, Regression, Cox; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.76 to 1.26]

3. Secondary Outcome: Number of Recurrent Episodes of VT or VF Requiring Antitachycardia Pacing (ATP) or ICD Shock Therapies
Description: Total number of recurrent ICD therapies requiring antitachycardia pacing (ATP) or shock will be analyzed, not just first event
Time Frame: 2 years of follow-up on average
Population: This outcome measure was an intent-to-treat analysis therefore all randomized subjects were included.
Measure: Count of Units; unit: VT/VF events
Units Other Than Participants: VT/VF events
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 510 | 502
Number analyzed (VT/VF events) | 741 | 986
VT/VF events | 433 | 650
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority; p = 0.028, Anderson-Gill analysis; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.51 to 0.96]

4. Secondary Outcome: Number of Patients With First Inappropriate ICD Shock
Description: Number of patients with first inappropriate ICD shock for other reasons than VT or VF
Time Frame: 2 years of follow-up on average
Population: This outcome measure was an intent-to-treat analysis therefore all randomized subjects were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 510 | 502
Participants | 16 | 20
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority; p = 0.398, Regression, Cox; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.38 to 1.47]

5. Secondary Outcome: Number of Patients With Hospitalization for Cardiac Causes or Death, Whichever Occurred First.
Description: Number of patients with a composite endpoint of cardiovascular hospitalization or death, whichever occurred first.
Time Frame: 2 years of follow-up on average
Population: This outcome measure was an intent-to-treat analysis therefore all randomized subjects were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 510 | 502
Participants | 237 | 222
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority; p = 0.316, Regression, Cox; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.91 to 1.34]

6. Secondary Outcome: Number of Patients With Heart Failure Hospitalization or Death, Whichever Occurred First
Description: Number of patients with a composite endpoint of heart failure hospitalization or death, whichever occurred first.
Time Frame: 2 years of follow-up on average
Population: This outcome measure was an intent-to-treat analysis therefore all randomized subjects were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 510 | 502
Participants | 144 | 140
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority; p = 0.577, Regression, Cox; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.84 to 1.37]

7. Secondary Outcome: Death
Description: Death as a safety endpoint of the trial
Time Frame: 2 years of follow-up on average
Population: This outcome measure was an intent-to-treat analysis therefore all randomized subjects were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 510 | 502
Participants | 70 | 78
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority; p = 0.871, Regression, Cox; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.69 to 1.37]

8. Secondary Outcome: Mean Meters Walked in 6 Minutes
Description: Exercise capacity measured by the 6-minute walk test
Time Frame: 1 year of follow-up
Population: Data was not collected on 86 patients in the placebo arm and 99 patients in the Ranolazine arm.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 325 | 353
meters | 314 (127.5) | 309 (123.5)
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority; p = 0.508, nonparametric Wilcoxon rank-sum test

9. Secondary Outcome: Quality of Life Measured by the Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a new, self-administered, 23-item questionnaire that quantifies physical limitations, symptoms, self-efficacy, social interference and quality of life. The scale ranges from 0-100 with lower scores indicating worse outcomes.
Time Frame: 1 year follow-up
Population: Data was not collected in 42 patients in the placebo arm and 61 patients in the Ranolazine arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 363 | 397
units on a scale | 73.6 (24.1) | 72.8 (24.3)
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority; p = 0.948, nonparametric Wilcoxon rank-sum test

10. Other Pre Specified Outcome: Number of Patients Whose First VT/VF Required Antitachycardia Pacing (ATP)
Description: Number of patients whose first VT or VF required antitachycardia pacing (ATP)
Time Frame: 2 years of follow-up on average
Population: This outcome measure was an intent-to-treat analysis therefore all randomized subjects were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 510 | 502
Participants | 92 | 117
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority; p = 0.038, Regression, Cox; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.55 to 0.98]

11. Other Pre Specified Outcome: Number of Patients Whose First VT/VF Required ICD Shock
Description: number of patients whose first VT or VF required ICD shock
Time Frame: 2 years of follow-up on average
Population: This outcome measure was an intent-to-treat analysis therefore all randomized subjects were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 510 | 502
Participants | 79 | 84
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority; p = 0.947, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.73 to 1.41]

12. Secondary Outcome: Number of Recurrent Inappropriate ICD Shocks
Description: Number of recurrent inappropriate ICD shocks in all patients combined.
Time Frame: 2 years of follow-up on average
Population: This outcome measure was an intent-to-treat analysis therefore all randomized subjects were included.
Measure: Number; unit: events
Arm/Group | Ranolazine | Placebo
Number analyzed (Participants) | 510 | 502
events | 19 | 26
Statistical Analysis 1: Comparison: Ranolazine vs Placebo; Test type: Superiority; p = 0.414, Anderdon-Gill analysis; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.36 to 1.52]

ADVERSE EVENTS:
Time Frame: approximately 2 years (median 27 months).
Arm/Group | Ranolazine | Placebo
All-Cause Mortality (participants affected / at risk) | 70/510 | 78/502
Serious Adverse Events (participants affected / at risk) | 0/510 | 0/502
Other Adverse Events (participants affected / at risk) | 69/510 | 17/502
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranolazine (N=510) | Placebo (N=502)
dizziness (General disorders) | 39 | 11
nausea (Gastrointestinal disorders) | 30 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2014-09-05): https://cdn.clinicaltrials.gov/large-docs/53/NCT01215253/Prot_000.pdf
  • Statistical Analysis Plan (2017-01-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT01215253/SAP_001.pdf